CLINICAL TRIAL: NCT01079871
Title: Evaluation of FID 114657 in Sjogren's Syndrome Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-65
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; Dry Eye
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FID 114657 (ORB Preserved Ocular Emulsion) (Experimental): ORB Preserved Ocular Emulsion dosed as needed throughout the day (PRN)
  Interventions: Other: FID 114657 (ORB Preserved Ocular Emulsion)

INTERVENTIONS:
Other: FID 114657 (ORB Preserved Ocular Emulsion) — Patients will dose as needed throughout the day (PRN) for 4 weeks.

SUMMARY:
The primary objective of this study is to assess the overall Sjogren's Syndrome subject's preference for a particular product. Dry eye symptom relief will also be evaluated based on clinical evaluation and a set of subject questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age, must read and sign the informed consent form (ICF), and must agree to comply with the study requirements.
* Patients must have a best corrected visual acuity of 0.6 LogMar or better in each eye, must report having an ocular examination in the last two years and must be using topical ocular dry eye therapy (artificial tears or Restasis) at least 4 times per day.
* Patients must have been diagnosed with Sjogren's Syndrome (confirmed or consistent with the American-European Consensus Criteria 2002).

Exclusion Criteria:

* Patients cannot wear contact lenses within one week prior to visit 1 and cannot wear their contact lenses during the study.
* Patients cannot have a history of hypersensitivity to any component of FID 114657, and cannot have diabetes (Type 1 or 2).
* Patients cannot have ocular or intraocular surgery or serious ocular trauma within the past 6 months, and cannot have an eyelid abnormality that might affect lid function.
* Patients cannot have punctal plugs that were placed less than or equal to 30 days prior to Visit 1, and cannot have active infections or inflammations not associated with Sjogren's Syndrome.
* They cannot have started or changed the dose of chronic systemic medication within 7 days prior to visit 1, and must remain on a stable dosing regimen for the duration of the study.
* Patients cannot have participated in another investigational clinical or research study within 30 days of visit 1 and are not allowed to participate in any other drug or device clinical trial for the duration of this study.
* Patients cannot have any findings in the vitreous, retina, macula and choroid that show signs of active inflammation and/or any structural change that in the opinion of the investigator is considered abnormal or unstable for that participant and/or a score of greater than 0 for the optic nerve.
* Patients can not have had punctal cauterization within 30 days prior to Visit 1, have a history of undergoing prior cataract surgery with complications as a result of the cataract surgery.
* Participants who have undergone prior cataract surgery without complications must be at least six months post-op with a stable refractive error.
* Patients cannot have received ocular prescription therapy in the last 30 days (Restasis can be used as long as stable for at least 30 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Preference based on subject's relief of dry eye | 5 weeks